CLINICAL TRIAL: NCT06359132
Title: The Effect of Integrated Mobile Health-supported Heart Rhythm Management Around Electrical Cardioversion in Terms of Cancelling Unnecessary Scheduled ECV Appointments in Patients With Presumed Persistent Atrial Fibrillation (TeleConvert-AF)
Brief Title: mHealth Rhythm Management in Terms of Cancelling Unnecessary Scheduled ECVs in Presumed Persistent AFpatients.
Acronym: TeleConvert-AF
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: TeleConvert-AF
Record Dates: First submitted 2024-01-09; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Arrhythmia; Mobile Health; Electrical Cardioversion
Keywords: Atrial fibrillation; Arrhythmia; Mobile health; Electrical cardioversion
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TeleConvert-AF: Patients with presumed persistent AF, age ≥18 years, scheduled for ECV, and in possession of a smartphone will be included in this study from January 2022 to January 2025.

SUMMARY:
Despite a clear definition in the European Society of Cardiology (ESC) guidelines, the differentiation between paroxysmal (self-terminating) and persistent (nonself- terminating) atrial fibrillation (AF) remains challenging in clinical practice. Some patients with presumed persistent AF are planned for electrical cardioversion (ECV) but appear to have a paroxysmal pattern or present in sinus rhythm (SR) at the scheduled ECV appointment. This results in unnecessary visits or interventions for patients, and costs and burden for the hospitals and health insurances. Based on the feasibility of the TeleCheck-AF approach, which is an on-demand mobile health (mHealth) infrastructure incorporating app-based heart rate and rhythm monitoring to support remote AF management through teleconsultation, the investigators aim to extend this mHealth approach to the management of presumed persistent AF patients planned for ECV.

DETAILED DESCRIPTION:
When putted on the waiting list for ECV (at baseline), the case-coordinator (investigator or nurse) will contact the patient and provide an mHealthprescription, manual and app-activation QR-code to use the CE-marked mobile phone app using photoplethysmography (PPG) technology through the built-in mobile phone's camera to monitor rate and rhythm. After 24-hours the case-coordinator will check whether the patient activated the app, otherwise will contact patient for further support.

Recordings from the device will be sent to a secure cloud application. This cloud application is equipped with an automatic analyses algorithm with a red-amber-green alert system. Patients will be asked to use the app 3-times a day and in case of symptom onset and disappearance while being on the waiting list for ECV. In case of amber alert (recording in asystole > 5 sec, tachycardia > 170 bpm, bradycardia 110 bpm) the subject's care team will be notified of the alert by the investigators within one workday. The subject will then be contacted by the care team to intensify rate control if necessary. Subjects also have the possibility to contact the investigators directly if needed. In case of green alert (SR recording), the investigators will process the alert within one workweek. The subject will then be contacted by the investigators to visit the hospital and execute a 12-lead ECG to confirm SR as soon as possible. When SR is confirmed by ECG, scheduled ECV will be cancelled by the treating physician and rate/rhythm control medication might be intensified, this is part of standard care. When SR is not confirmed by ECG, treatment decisions will remain to the treating physician and he/she will decide whether or not to cancel scheduled ECV (based on PPG recordings). In the 4-weeks following scheduled ECV appointment, all patients will receive remote semi-continuous app-based rate/rhythm monitoring including red-amber- green alert notifications and will be asked to use the app 3-times a day and in case of symptom onset and disappearance. In case of an amber alert, the subject's care team will be notified of the alert by the investigators within one workday. The subject will then be contacted by the care team to intensify rate control if necessary. Subjects also have the possibility to contact the investigators directly if needed. Of importance is that alerts will only be assessed by the investigators during office hours. Patients will specifically (both verbally and written) be informed that in case of alarming symptoms during or outside of office hours, emergency services or their own general practitioner should be contacted. In all cases of acute emergencies, a patient should contact the emergency services. Furthermore, patients will be asked to fulfill a self-composed questionnaire based on the System Usability Scale extended with additional questions to assess the usability and user-friendliness of the refined TeleCheck-AF approach around ECV at 4-week follow-up. Also a self-composed questionnaire based on the HADS-A scale will be used to assess anxiety while using the mHealth-based refined TeleCheck-AF approach around ECV at four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Presumed persistent AF
* Scheduled for ECV
* Age ≥18 years
* Smartphone possession
* Ability and willing to sign informed consent
* Ability and willing to use mobile phone app (FibriCheck)

Exclusion Criteria:

* Deemed unsuitable for participation by attending physician
* Presence of an active implanted electronic cardiac device

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with presumed persistent AF, age ≥18 years, scheduled for ECV, and in possession of a smartphone will be included in this study from January 2022 to January 2024.
Sampling Method: Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The number of cancelled unnecessary scheduled ECV appointments in patients with presumed persistent AF scheduled for ECV unnecessary scheduled ECV appointments | through study completion, an average of 8 weeks
  The number of cancelled unnecessary scheduled ECV appointments in patients with presumed persistent AF scheduled for ECV

SECONDARY OUTCOMES:
Number of patients that agreed the refined TeleCheck-AF approach is usable and userfriendly as assessed by the System Usability Scale questionnaire extended with additional questions | through study completion, an average of 8 weeks
  Number of patients that agreed the refined TeleCheck-AF approach is usable and userfriendly as assessed by the System Usability Scale questionnaire extended with additional questions
Number of patients that agreed the refined TeleCheck-AF approach is anxious as assessed by the HADS-A scale questionnaire | through study completion, an average of 8 weeks
  Number of patients that agreed the refined TeleCheck-AF approach is anxious as assessed by the HADS-A scale questionnaire
Amount of saved costs for the hospitals and health insurances by using the TeleCheck-AF approach preceding ECV in terms of cancelling unnecessary scheduled ECV appointments | through study completion, an average of 8 weeks
  Amount of saved costs for the hospitals and health insurances by using the TeleCheck-AF approach preceding ECV in terms of cancelling unnecessary scheduled ECV appointments
Number of patients with paroxysmal AF | through study completion, an average of 8 weeks
  Number of patients with paroxysmal AF assessed by the refined by the on-demand heart rate and rhythm monitoring application
Time to recurrence of AF | up to 4 weeks after ECV
  Time to recurrence of AF
Time period of monitoring heart rate and rhythm using the mHealth-based application | through study completion, an average of 8 weeks
  Time period of monitoring heart rate and rhythm using the mHealth-based application
Amount of burden for the hospitals and health insurances by using the TeleCheck-AF approach preceding ECV in terms of cancelling unnecessary scheduled ECV appointments | through study completion, an average of 8 weeks
  Amount of burden for the hospitals and health insurances by using the TeleCheck-AF approach preceding ECV in terms of cancelling unnecessary scheduled ECV appointments

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Viecuri Medical Center, Venlo, Limburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engels MDEA, Hermans ANL, Hermans BJM, Luermans J, Chaldoupi SM, Hendriks JML, Lankveld T, Kessels MVM, Vorstermans BJGH, Beukema RJ, Vernooy K, Heesen W, Linz DK. Smartphone application-based heart rhythm monitoring to cancel scheduled electrical cardioversion in patients with spontaneous conversion of presumed persistent atrial fibrillation: TeleConvert-AF. Eur Heart J Digit Health. 2025 Dec 9;7(2):ztaf140. doi: 10.1093/ehjdh/ztaf140. eCollection 2026 Mar. PMID 41624561